CLINICAL TRIAL: NCT06438757
Title: Phase IIa Trial to Evaluate the Pharmacokinetic/Pharmacodynamic Characteristics and Safety of JYB1904 in Patients With Allergic Asthma
Brief Title: Trial of JYB1904 in Patients With Allergic Asthma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYB1904-201
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JYB1904: Dose-1 (Experimental)
  Interventions: Drug: JYB1904
- JYB1904: Dose-2 (Experimental)
  Interventions: Drug: JYB1904
- JYB1904: Dose-3 (Experimental)
  Interventions: Drug: JYB1904
- Omalizumab (Active Comparator)
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: JYB1904 — Participants will receive JYB1904 every 8 weeks for 24 weeks.
  Arms: JYB1904: Dose-1; JYB1904: Dose-2; JYB1904: Dose-3
Drug: Omalizumab — Participants will receive Omalizumab every 2/4 weeks for 24 weeks.
  Arms: Omalizumab

SUMMARY:
This phase IIa trial is meant to evaluate the pharmacokinetics, pharmacodynamics and safety of JYB1904 in patients with allergic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent voluntarily;
* Aged 18-75 years, weight ≥ 40 kg, male or female;
* Diagnosed Allergic asthma.

Exclusion Criteria:

* Prior exposure to anti-IgE therapy within 1 year;
* Allergic to anti-IgE biologics;
* Current smokers, or quit smoking within 1 year;
* Combined with other non-allergic diseases that cause IgE elevation；
* History of malignancy, autoimmune diseases, Immune complex mediated diseases, Hypereosinophilic syndrome;
* Other conditions unsuitable for the trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Serum concentrations of JYB1904 | Baseline through 337 days post-dose
  Serum concentrations of JYB1904, assessed by pre-specified methods
Serum concentrations of IgE | Baseline through 337 days post-dose
  Serum concentrations of IgE, assessed by pre-specified methods
Adverse Events(AEs) | Baseline through 337 days post-dose
  Incidence and features of AEs assessed by CTCAE v5.0, and related safety parameters analysis

SECONDARY OUTCOMES:
Times of protocol-defined asthma exacerbations during the 24-week treatment period | Baseline through 168 days post-dose
  Times of protocol-defined asthma exacerbations during the 24-week treatment period
Change in spirometry measures of forced expiratory volume in one second (FEV1) in 24 weeks | Baseline through 24 weeks post-dose
  forced expiratory volume in one second (FEV1)
Serum concentrations of anti-drug antibody (ADA) | Baseline through 337 days post-dose
  Serum ADA assessed by pre-specified methods, and related immunogenic features analysis

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhang, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China